CLINICAL TRIAL: NCT00818077
Title: Using Continuous Glucose Monitoring to Understand the Glycemic Impact of Food
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: 03654-07-A
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes; Currently Taking Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metformin, Type 2 Diabetes
  Interventions: Other: Continuous Glucose Monitoring of Carbohydrate Intake

INTERVENTIONS:
Other: Continuous Glucose Monitoring of Carbohydrate Intake — Subjects eat standard breakfast and lunch and keep food records.
  Other Names: Navigator CGM System

SUMMARY:
This study will look at the impact that meals have on blood glucose (sugar) levels. Subjects will be asked to use a Continuous Glucose Monitoring System (CGM), which monitors glucose levels continuously. Breakfast and lunch meals will be provided and must be consumed at the International Diabetes Center.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* Age 18 and older
* Diagnosed with type 2 diabetes for a minimum of 6 months
* Is taking metformin for diabetes management; no other diabetes medications
* Has been on a stable dose of metformin for at least 3 months
* HbA1c is 7% or greater and less than 9%; >7% or <9%
* BMI <30kg/m2
* Willing to give informed consent
* No evidence of acute illness, fever, undue stress
* Motivated and capable of following the protocol and instructions provided by the healthcare professional
* Available for the study on the scheduled visit days
* Access to telephone communications

Exclusion Criteria:

* Under 18 years of age
* Has not been diagnosed with type 2 diabetes for a minimum of 6 months
* Is currently taking other diabetes medications in addition to metformin
* Has taken other diabetes medications within the past 3 months
* HbA1c <7% or >9%
* BMI > 30kg/m2
* Unable to follow the study protocol
* No access to telephone communications
* Unable to read and write in English
* Unable to maintain their health, or have undue stress
* Skin abnormalities at the insertion sites that would confound assessment of the effect of the device on the skin
* Allergy to adhesives
* Any concomitant medical condition that would likely affect the evaluation of device performance
* Taken oral or inhaled prednisone or cortisone medications in the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes, 18 years of age of older, currently taking metformin
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Glycemic Response to the Fixed Meal | 4 hour meal test

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Powers, PhD, RD, CDE, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] American Diabetes Association. Nutrition Recommendations and Interventions for Diabetes: a position statement of the American Diabetes Association. Diabetes Care. 2007 Jan;30 Suppl 1:S48-65. doi: 10.2337/dc07-S048. No abstract available. PMID 17192379
- [Background] Franz MJ, Boucher JL, Green-Pastors J, Powers MA. Evidence-based nutrition practice guidelines for diabetes and scope and standards of practice. J Am Diet Assoc. 2008 Apr;108(4 Suppl 1):S52-8. doi: 10.1016/j.jada.2008.01.021. PMID 18358257
- [Background] Crapo PA, Reaven G, Olefsky J. Postprandial plasma-glucose and -insulin responses to different complex carbohydrates. Diabetes. 1977 Dec;26(12):1178-83. doi: 10.2337/diab.26.12.1178. PMID 590639